CLINICAL TRIAL: NCT02353780
Title: Mechanistic Studies of B- and T-Cell Function in Rheumatoid Arthritis Patients Treated With TNF Antagonists, Tocilizumab, or Abatacept
Brief Title: Mechanistic Studies of B- and T-Cell Function in RA Patients Treated With TNF Antagonists, Tocilizumab, or Abatacept
Acronym: MAZERATI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Dr. Larry W. Moreland (Other)
Collaborators: Genentech, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Dr. Larry W. Moreland, Chief, Division of Rheumatology and Clinical Immunology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY19040127
Record Dates: First submitted 2013-06-30; First posted 2015-02-03 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid arthritis; TNF inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tumor Necrosis Factor Inhibitors; Etanercept; Infliximab; Certolizumab Pegol; Adalimumab; Abatacept; tocilizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Different TNF inhibitor (Active Comparator): The participant will be prescribed any TNF antagonist in this arm. The treating rheumatologist selects the TNF antagonist and the appropriate options for that therapy.
  Interventions: Drug: TNF Antagonist (enbrel, humire, remicade, cimzia, symponi)
- Abatacept (Active Comparator): The participant will be prescribed abatacept in this arm. The treating rheumatologist selects the appropriate options for that therapy.
  Interventions: Drug: Abatacept
- Tocilizumab (Active Comparator): The participant will be prescribed tocilizumab. The treating rheumatologist selects the appropriate options for that therapy.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: TNF Antagonist (enbrel, humire, remicade, cimzia, symponi) — TNF Antagonist; treating rheumatologist selects specifics for the therapy chosen.
  Other Names: Enbrel; Humira; Remicade; Cimzia; Symponi
  Arms: Different TNF inhibitor
Drug: Abatacept — Abatacept; SQ; specifics to be determined by the treating rheumatologist.
  Other Names: Orencia
  Arms: Abatacept
Drug: Tocilizumab — Tocilizumab; SQ; specifics determined by the treating rheumatologist.
  Other Names: Actemra
  Arms: Tocilizumab

SUMMARY:
An Agency for Healthcare Research and Quality executive summary indicated that better comparative effectiveness trial designs are needed to determine the relative merits of existing versus new and expensive biologic drug therapies for rheumatoid arthritis (RA). There are now 9 biologic therapies approved for treating RA. Four classes of biologics (TNF antagonists, B-cell inhibitors, T-cell co-stimulator blocker, and Interleukin-6 receptor blocker) are approved for use in RA patients with moderate or severe disease activity. Several critical questions have arisen, such as 1) what therapy should be prescribed after failure of methotrexate and/or other oral disease modifying antirheumatic drugs (DMARDs) to adequately control disease activity; 2) what is the level of efficacy of the various biologic therapies when compared in head-to-head trials; and 3) what are the mechanisms associated with failure of methotrexate and/or other oral DMARD therapy and responsiveness to biologic therapies. The MAZERATI study will provide the foundation for answering these questions and determining the mechanisms associated with these biologic therapies.

DETAILED DESCRIPTION:
Single center, randomized, assessor-blinded, observational longitudinal assessment. Subjects will be randomized to treatment with an anti-TNF therapy, tocilizumab or abatacept and evaluated at baseline, and after 1, 3 and 6 months of therapy. All biologics will be administered subcutaneously (SQ). A blinded assessor will perform clinical disease activity assessments and blood samples will be obtained for mechanistic studies.

After randomization, patients must take at least one dose of the assigned medication and must maintain their baseline prednisone and oral disease modifying anti-rheumatic drug (DMARD) medications until they have received their first dose of assigned medication to be considered per protocol participants. During the first 3 months of therapy, patients and their physicians will be permitted to taper but not increase corticosteroids. Adjustments of study medication or oral DMARDs will not be permitted during the first 3 months of the study except as outlined in the protocol. Adjustments or additions of analgesics will be permitted throughout the study period.

Following randomization and treatment initiation, study participants will be seen in the clinic at 1 month (3-5 weeks), 3 months (10-14 weeks), and 6 months (22-30 weeks) after the initiation of therapy; at each time point, a blinded clinical disease activity assessment will occur and blood samples will be obtained for mechanistic studies. The occurrence and severity of unanticipated problems will be recorded continuously throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA by a physician as defined by the 1987 and/or 2010 ACR criteria.
* 18 years of age or less than or equal to 64 at the time of diagnosis of RA.
* RA Disease Activity CDAI > 10
* If using oral corticosteroids, must have been on stable dose (≤ 10 mg/day) for at least 2 weeks prior to study drug initiation.
* PPD negative or if PPD positive documentation of therapy with INH for at least 1 month prior to study initiation and negative chest x-ray.
* Must have been treated within the past year with either methotrexate (MTX), leflunomide (LEF), hydrochloroquine (HCQ) and/or sulfasalazine (SSZ) for ≥ 3 months.
* Prior or concurrent use of other oral DMARD therapy, including MTX, leflunomide, SSZ, and HCQ, is permitted. Patients taking oral DMARDs must be on stable doses of DMARDs for at least 4 weeks prior to study drug initiation. Subjects are not required to be taking an oral DMARD.

Exclusion Criteria:

* Use of cyclophosphamide, penicillamine, cyclosporine A, tacrolimus or gold therapy is not permitted in the 6 months prior to enrollment.
* Patients who are using or have used other biologic agents or tofacitinib concomitantly or prior to this study
* History of active and/or chronic infection such as hepatitis, pneumonia, pyelonephritis,herpetic infections or chronic skin infections and any active opportunistic infection, including but not limited to evidence of active cytomegalovirus, active Pneumocystis carinii, aspergillosis, histoplasmosis or atypical mycobacterium infection.
* Active TB or evidence of latent TB (positive PPD skin test or a history of old or latent TB on chest x-ray) without adequate therapy for TB.
* Pregnant or lactating women.
* Patients with current signs or symptoms of uncontrolled renal, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
* Diagnosis of liver disease or elevated hepatic enzymes, as defined by ALT, AST or both >1.5 x the upper limit of normal (ULN) or total bilirubin > ULN.
* Any of the following hematologic abnormalities, confirmed by repeat tests:

  1. White blood count < 3,000/µL or > 14,000/µL
  2. Lymphocyte count <500/µL
  3. Platelet count < 100,000/µL
  4. Hemoglobin < 8.0 g/dL
  5. Neutrophil count < 2,000 cells/µL
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Immunization with a live/attenuated vaccine within 2 months prior to baseline or 3 months of last study visit.
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Patients with reproductive potential not willing to use an effective method of contraception
* History of alcohol, drug or chemical abuse with 1 year prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry W. Moreland, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 10 enrolled subjects, 9 subjects were randomized to one of three arms. One subject withdrew consent prior to being screened/randomized.
Period: Overall Study
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Full Range); unit: years] | 44 [25 to 60] | 51 [43 to 60] | 52 [42 to 61] | 49 [25 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 0 | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
CDAI [Mean (Full Range); unit: units on a scale] — Clinical Disease Activity Index (CDAI) is a composite score of RA disease activity based on patient survey (up to 10 points), physician survey (up to 10 points), + number of swollen joints + number of tender joints. 0 = no disease, max score is 60, higher score = more severe disease.
  units on a scale | 23 [10.5 to 30] | 17.3 [6.5 to 27.5] | 17.3 [14 to 20] | 19.2 [6.5 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Mechanistic Comparisons (Changes in Frequencies of Peripheral Blood Immune Cell Subsets Following Institution of a Subcutaneously Administered TNF Antagonist, Tocilizumab or Abatacept.)
Description: There will be no primary efficacy endpoints for the study. The primary endpoint of the study will be changes in frequencies of peripheral blood immune cell subsets following institution of a subcutaneously administered TNF antagonist, tocilizumab or abatacept. Flow ctyometry was performed on peripheral blood T cells to determine frequency of Th17/TfH cells based on cell surface markers.
Time Frame: 0 to 3 months
Population: Patients (total of 5) who provided blood samples at 0 and 3 months and flow cytometry was performed before study discontinuation are included in the analysis.
Measure: Mean (Full Range); unit: Th17/TfH cell subset % change
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 2 | 1 | 2
Th17/TfH cell subset % change | 0.9 [0.38 to 1.46] | 2.9 [2.9 to 2.9] | 0.9 [0.7 to 1.1]

2. Secondary Outcome: Efficacy (CDAI)
Description: Efficacy of therapy, as measured by number of participants with Clinical Disease Activity Index (CDAI) of less than 2.8 (remission). CDAI is a composite score of RA disease activity based on patient survey (up to 10 points), physician survey (up to 10 points), + number of swollen joints + number of tender joints. 0 = no disease, max score is 60, higher score = more severe disease. Number of patients achieving remission is reported.
Time Frame: 0 to 3 months
Population: CDAI change from 0 to 3 months was calculated for the 5 patients who had this data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 2 | 1 | 2
Participants | 0 | 0 | 0

3. Secondary Outcome: Efficacy (DAS)
Description: Efficacy as measured by DAS remission with a DAS28-CRP < 2.4
Time Frame: 3 month and 6 month
Population: CRP assays were not run as the study was incomplete due to premature termination of study.
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: ACR20, 50, and 70 Response
Description: Efficacy as measured by ACR20, 50, and 70 response at 3 months and 6 months versus baseline
Time Frame: 3 month and 6 month
Population: ACR20, 50, 70 were not calculated since clinical parameter such as CRP were not collected due to premature termination of study.
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Efficacy (EULAR)
Description: Efficacy as measured by European League against rheumatism (EULAR) response
Time Frame: 3 month and 6 month
Population: This parameter was not calculated as data was incomplete due to premature termination of study
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Adherence
Description: Adherence to drug regimen over course of clinical study
Time Frame: 3 month and 6 month
Population: Number of patients who adhered to drug treatment through 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 3 | 3 | 3
Participants | 3 | 3 | 3

7. Secondary Outcome: Steroid Use
Description: Number of patients with steroid doses remaining below 10 mg/day
Time Frame: 3 month and 6 month
Population: Steroid dose information was not collected at 3 and 6 months as the study was terminated early with insufficient patient enrollment.
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Corticosteroid Use
Description: Average corticosteroid dose
Time Frame: 3 month and 6 month
Population: Data not collected due to early termination of study
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: DMARD Use
Description: Number of patients without additional oral DMARDs or with a reduction in the number of oral DMARDs
Time Frame: 3 month and 6 month
Population: Data was not collected for DMARDs due to premature termination of study due to insufficient patient enrollment.
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Reason for Discontinuation of Treatment
Description: Reason for discontinuation of treatment as provided by patient/provider (side effects, lack of efficacy, cost, patient compliance, etc.)
Time Frame: 3 month and 6 month
Population: all 9 patients enrolled and assigned to a study group were analyzed for completion of therapy. All patients completed therapy and none discontinued so no additional data to report.
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of study participation which was 6 months.
Arm/Group | Different TNF Inhibitor | Abatacept | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Different TNF Inhibitor (N=3) | Abatacept (N=3) | Tocilizumab (N=3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Increase in cholesterol levels (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Eye floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the small number of patients enrolled in each group, it was not possible to perform statistical analyses of the primary endpoints. These are fairly broad measures that require large numbers to identify patterns in subset changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02353780/Prot_SAP_000.pdf